CLINICAL TRIAL: NCT04784442
Title: A Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group Trial to Evaluate the Efficacy and Safety of ETC-1002 in Patients With Hypercholesterolemia
Brief Title: A Dose-finding Trial of ETC-1002(Bempedoic Acid) in Patients With Hypercholesterolemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 346-102-00001; jRCT2031200445 (Other: jRCT)
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Results first posted 2024-03-04 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- ETC-1002 180mg (Experimental)
  Interventions: Drug: 180mg of ETC-1002(bempedoic acid)
- ETC-1002 120mg (Experimental)
  Interventions: Drug: 120mg of ETC-1002(bempedoic acid)
- ETC-1002 60mg (Experimental)
  Interventions: Drug: 60mg of ETC-1002(bempedoic acid)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: 180mg of ETC-1002(bempedoic acid) — 180mg, tablet, once daily, for 12 weeks
  Arms: ETC-1002 180mg
Drug: 120mg of ETC-1002(bempedoic acid) — 120mg, tablet, once daily, for 12 weeks
  Arms: ETC-1002 120mg
Drug: 60mg of ETC-1002(bempedoic acid) — 60mg, tablet, once daily, for 12 weeks
  Arms: ETC-1002 60mg
Drug: Placebo — placebo, tablet, once daily, for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to assess the low-density lipoprotein cholesterol (LDL-C)-lowering efficacy and safety of ETC-1002(bempedoic acid) 60 mg, 120 mg and 180 mg versus placebo added to ongoing stable statin therapy or other lipid-modifying therapies in Japanese patients with hypercholesterolemia treated for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have obtained informed consent to all of the observation/examination/evaluation items specified in the protocol
* Patients must be on stable statin therapy defined as atorvastatin, pitavastatin, rosuvastatin, pravastatin, simvastatin, or fluvastatin daily[and other lipid-modifying therapies(LMTs) if needed] at least 4 weeks(6 weeks for fibrates) prior to screening and above LDL-C control target. Or Patients for statin intolerant must be on stable LMT(s) at least 4 weeks prior to screening and above LDL-C control target. Statin intolerance defined as an inability to tolerate 1 or more statins due to an adverse safety effect that started or increased during statin therapy and resolved or improved when statin therapy was discontinued or decreased. Patients on the lowest or under the dosage of the approved dose of statin or unable to tolerate any statin at any dose were eligible. Patients could continue taking the lowest or under the dosage of the approved dose of statin therapy or taking other LMTs throughout the study provided that it was stable and well tolerated.
* Fasting mean TG level < 400 mg/dL from measurements at screening
* Other protocol specific inclusion criteria may apply

Exclusion Criteria:

* Women who are pregnant or breastfeeding or who have a positive pregnancy test (urine) result at screening or baseline visits
* Sexually active male subjects or sexually active female subjects of childbearing potential who do not agree to practice 2 different methods of birth control or to remain abstinent during the trial and for 30 days after final IMP administration test (urine) result at screening or baseline visits
* Patients with homozygous familial hypercholesterolemia (HoFH)
* Patients with a history or current symptoms of any of the following clinically significant cardiovascular diseases within 3 months prior to screening or before baseline visit

  * Myocardial infarction, severe or unstable angina pectoris, coronary angioplasty, coronary artery bypass graft, stroke, transient ischemic attack, symptomatic carotid artery stenosis, symptomatic peripheral arterial disease, or decompensated heart failure
  * Abdominal aortic aneurysm
  * Unexplained syncope or long-QT syndrome, family history of long-QT syndrome, or risk factors for Torsade de Pointes, such as persistent hypokalemia or second- or third-degree atrioventricular block (except when controlled by medication, etc)
* Uncontrolled hypertension, defined as follows:

  * Sitting systolic blood pressure after resting 5 minutes of ≥160 mmHg or diastolic blood pressure of ≥100 mmHg at screening
* Patients with uncontrolled and serious hematologic or coagulation disorders or with Hgb of <10.0 g/dL at screening
* Patients with type 1 diabetes or uncontrolled type 2 diabetes with hemoglobin A1c (HbA1c) of ≥9% at screening
* Patients with uncontrolled hypothyroidism with thyroid-stimulating hormone (TSH) of >1.5 × ULN at screening
* Patients with liver disease or dysfunction, including:

  * Positive serology for hepatitis B surface antigen (HBsAg) and/or hepatitis C antibodies at screening
  * Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) of ≥3 × ULN and/or total bilirubin of ≥2 × ULN
* Patients with creatine kinase (CK) elevation( >3 × ULN) at screening
* Patients with renal dysfunction or nephritic syndrome or a history of nephritis and with estimated glomerular filtration rate (eGFR) of ≤30 mL/min/1.73m2 at screening
* Other protocol specific inclusion criteria may apply

Ages: 20 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2021-03-24 (Actual); Primary Completion 2022-04-18 (Actual); Study Completion 2022-05-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Takehisa Matsumaru, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (1):
- Tokyo-Eki Center-Building Clinic, Chuo-ku,Tokyo, Japan

IPD SHARING:
Plan to Share IPD: Yes
: Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal.
Supporting Information: Study Protocol, SAP
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article Publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com.

RESULTS

PARTICIPANT FLOW:
Groups:
- ETC-1002 60 mg: ETC-1002 60 mg tablet once daily for 12 weeks.
- ETC-1002 120 mg: ETC-1002 120 mg tablet once daily for 12 weeks.
- ETC-1002 180 mg: ETC-1002 180 mg tablet once daily for 12 weeks.
- Placebo: Placebo tablet once daily for 12 weeks.
Period: Overall Study
Arm/Group | ETC-1002 60 mg | ETC-1002 120 mg | ETC-1002 180 mg | Placebo
Started | 47 | 46 | 48 | 47
Completed | 44 | 46 | 46 | 46
Not Completed | 3 | 0 | 2 | 1
Not completed — Adverse Event | 1 | 0 | 2 | 1
Not completed — Protocol Violation | 1 | 0 | 0 | 0
Not completed — Non-compliance with study drug | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: For the full analysis set (FAS), a total of 186 subjects (45 for the 60 mg group, 46 for the 120 mg group, and 48 for the 180 mg group were included in the ETC-1002 group, and 47 subjects were included in the placebo group).
Groups:
- Total: Total of all reporting groups
Arm/Group | ETC-1002 60 mg | ETC-1002 120 mg | ETC-1002 180 mg | Placebo | Total
Number analyzed (Participants) | 45 | 46 | 48 | 47 | 186
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0 | 0
  Between 18 and 65 years | 28 | 27 | 23 | 20 | 98
  >=65 years | 17 | 19 | 25 | 27 | 88
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.9 (9.26) | 60.4 (8.94) | 60.4 (11.98) | 63.0 (10.65) | 61.2 (10.28)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 16 | 12 | 60
  Male | 29 | 30 | 32 | 35 | 126
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 45 | 46 | 48 | 47 | 186
Region of Enrollment [Number; unit: participants]
  Japan | 45 | 46 | 48 | 47 | 186

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in LDL-C From Baseline to Week 12
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100. Baseline was defined as the mean of the values from Week -1 and Day 1. When LDL-C at Week 12 was missing, the missing value was imputed using the last observation carried forward from the start of the IMP administration to 2 days after the final IMP administration.
Time Frame: Baseline, week12
Population: The FAS included all subjects who receive at least one dose of IMP during the treatment period and for whom LDL-C values at baseline and at least one post-dose (up to 2 days after final IMP administration) are observed.
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 60 mg | ETC-1002 120 mg | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 45 | 46 | 48 | 47
Percent Change | -10.59 (2.153) | -21.85 (2.156) | -21.26 (2.095) | -1.92 (2.117)
Statistical Analysis 1: Comparison: ETC-1002 180 mg vs Placebo; Test type: Superiority — The overall Type I error rate will be controlled by performing comparison versus the placebo group starting from the highest ETC 1002 dose group by a closed testing procedure at a two-sided significance level of 0.05; p < 0.001, ANCOVA; Least squares mean difference = -19.35, 95% CI 2-sided [-24.81 to -13.88], Standard Error of Mean 2.768 — The least squares mean difference was calculated as the value for the ETC-1002 180 mg arm minus the value for the placebo arm
Statistical Analysis 2: Comparison: ETC-1002 120 mg vs Placebo; Test type: Superiority; p < 0.001, ANCOVA; Least squares mean difference = -19.93, 95% CI 2-sided [-25.45 to -14.41], Standard Error of Mean 2.798 — The least squares mean difference was calculated as the value for the ETC-1002 120 mg arm minus the value for the placebo arm
Statistical Analysis 3: Comparison: ETC-1002 60 mg vs Placebo; Test type: Superiority; p = 0.002, ANCOVA; Least squares mean difference = -8.67, 95% CI 2-sided [-14.22 to -3.12], Standard Error of Mean 2.813; The least squares mean difference was calculated as the value for the ETC-1002 60 mg arm minus the value for the placebo arm

2. Secondary Outcome: Percent Change in HDL Cholesterol From Baseline to Week 12
Description: Percent change from Baseline was calculated as the ([post-Baseline value minus the Baseline value] divided by the Baseline value) x 100.
Time Frame: Baseline, week12
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 60 mg | ETC-1002 120 mg | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 45 | 46 | 48 | 47
Percent Change | 0.16 (2.208) | -0.65 (2.190) | -7.29 (2.139) | 3.08 (2.155)

3. Secondary Outcome: Percent Change in Non-HDL Cholesterol From Baseline to Week 12
Description: as for outcome 2
Time Frame: Baseline, week12
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 60 mg | ETC-1002 120 mg | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 45 | 46 | 48 | 47
Percent Change | -8.86 (2.019) | -18.29 (2.021) | -16.01 (1.956) | -1.62 (1.988)

4. Secondary Outcome: Percent Change in Total Cholesterol From Baseline to Week 12
Description: as for outcome 2
Time Frame: Baseline, week12
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 60 mg | ETC-1002 120 mg | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 45 | 46 | 48 | 47
Percent Change | -6.42 (1.665) | -13.61 (1.650) | -13.56 (1.599) | -0.55 (1.621)

5. Secondary Outcome: Percent Change in Triglycerides From Baseline to Week 12
Description: as for outcome 2
Time Frame: Baseline, week12
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 60 mg | ETC-1002 120 mg | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 45 | 46 | 46 | 47
Percent Change | -9.09 (6.286) | -5.62 (6.290) | 9.17 (6.151) | -0.08 (6.219)

6. Secondary Outcome: Percent Change in Apolipoprotein B From Baseline to Week 12
Description: as for outcome 2
Time Frame: Baseline, week12
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 60 mg | ETC-1002 120 mg | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 45 | 46 | 46 | 47
Percent Change | -8.18 (1.715) | -14.59 (1.709) | -12.47 (1.704) | -2.13 (1.704)

7. Secondary Outcome: Percent Change in High Sensitivity C Reactive Protein From Baseline to Week 12
Description: as for outcome 2
Time Frame: Baseline, week12
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 60 mg | ETC-1002 120 mg | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 45 | 46 | 46 | 47
Percent Change | 150.54 (62.494) | 1.02 (62.418) | -34.58 (62.745) | 0.98 (61.513)

8. Secondary Outcome: Percent Change in Hemoglobin A1c From Baseline to Week 12
Description: as for outcome 2
Time Frame: Baseline, week12
Measure: Least Squares Mean (Standard Error); unit: Percent Change
Arm/Group | ETC-1002 60 mg | ETC-1002 120 mg | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 45 | 46 | 46 | 47
Percent Change | 0.11 (0.591) | -0.40 (0.596) | -0.21 (0.592) | -0.05 (0.578)

9. Secondary Outcome: Proportion of Subjects Whose LDL-C Value Achieved the Lipid Management Goals Based on Risk Assessment at Week 12
Description: The proportion of subjects whose LDL-C value achieves the lipid management goal at Week 12.
Time Frame: Baseline, week12
Measure: Number; unit: participants
Arm/Group | ETC-1002 60 mg | ETC-1002 120 mg | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 45 | 46 | 48 | 47
participants | 15 | 26 | 28 | 1

10. Secondary Outcome: Proportion of Subjects Whose LDL-C Value Achieve < 70 mg/dL at Week 12
Description: The proportion of subjects whose LDL-C value achieves <70 mg/dL at Week 12.
Time Frame: Baseline, week12
Measure: Count of Participants; unit: Participants
Arm/Group | ETC-1002 60 mg | ETC-1002 120 mg | ETC-1002 180 mg | Placebo
Number analyzed (Participants) | 45 | 46 | 48 | 47
Participants | 0 | 1 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were monitored from signing of the informed consent form until follow-up for up to 28 (+7) days after the last dose of study medication.
Description: The safety analysis set will include subjects who receive at least one dose of IMP during the treatment period.
Arm/Group | ETC-1002 60 mg | ETC-1002 120 mg | ETC-1002 180 mg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/46 | 0/47 | 0/48
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/46 | 1/47 | 1/48
Other Adverse Events (participants affected / at risk) | 23/47 | 17/46 | 21/48 | 9/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ETC-1002 60 mg (N=47) | ETC-1002 120 mg (N=46) | ETC-1002 180 mg (N=47) | Placebo (N=48)
Dental cyst (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ETC-1002 60 mg (N=47) | ETC-1002 120 mg (N=46) | ETC-1002 180 mg (N=48) | Placebo (N=47)
Abdominal pain upper (Gastrointestinal disorders) | 4 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 3 | 1 | 1 | 1
Large intestine polyp (Gastrointestinal disorders) | 0 | 2 | 0 | 0
Fatigue (General disorders) | 2 | 1 | 1 | 0
Malaise (General disorders) | 1 | 3 | 3 | 0
Pyrexia (General disorders) | 5 | 4 | 1 | 2
Vaccination site pain (General disorders) | 1 | 3 | 0 | 1
Vaccination site swelling (General disorders) | 0 | 2 | 1 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 2 | 0 | 5 | 0
Nasopharyngitis (Infections and infestations) | 2 | 1 | 1 | 0
Otitis externa (Infections and infestations) | 0 | 2 | 0 | 0
Vaccination complication (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0
Alanine aminotransferase increased (Investigations) | 0 | 2 | 3 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 2 | 1
Blood creatine phosphokinase increased (Investigations) | 1 | 1 | 2 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 2 | 0
Blood uric acid increased (Investigations) | 2 | 3 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 2 | 3 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 2 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 2
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 2 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 0 | 5 | 2 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0 | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-11-19): https://cdn.clinicaltrials.gov/large-docs/42/NCT04784442/Prot_000.pdf
  • Statistical Analysis Plan (2022-06-20): https://cdn.clinicaltrials.gov/large-docs/42/NCT04784442/SAP_001.pdf